CLINICAL TRIAL: NCT04650152
Title: A Prospective Observational Study to Assess Tricor Therapy Effectiveness in Patients With Metabolic Syndrome (TRISTAN)
Brief Title: Study to Assess Tricor Therapy Effectiveness in Patients With Metabolic Syndrome (TRISTAN)
Acronym: TRISTAN
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: FENO5002
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Hypertriglyceridemia; Metabolic Syndrome
Keywords: Tricor; fenofibrate; metabolic syndrome; hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia; Metabolic Syndrome | interventions — Fenofibrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fenofibrate: Adult patients with triglycerides > 2,3 mmol/l who are on statins and who are primary prescribed fenofibrate (or fenofibrate treatment break is at least 6 months) in accordance with ordinary physician practice in Russia.
  Interventions: Drug: Tricor (fenofibrate), 145 mg, film-coated tablet

INTERVENTIONS:
Drug: Tricor (fenofibrate), 145 mg, film-coated tablet — Observational study without intervention. Fenofibrate is prescribed in routine manner in accordance with clinical practice and the valid Instruction for Medical Use regarding the dose, duration of therapy, patient population, and therapeutic indication.
  Other Names: Tricor

SUMMARY:
This study is a prospective observational program within the frames of which Tricor (fenofibrate) is prescribed to patients with hypertriglyceridemia within a routine procedure as a part of the combination therapy with statins.

DETAILED DESCRIPTION:
Metabolic syndrome is a cluster of interrelated risk factors that leads to metabolic dysregulation and atherosclerotic cardiovascular diseases. The increased risk of cardiovascular disease in people with metabolic syndrome has been well established by observational studies and meta-analyses.

Strategies to reduce cardiovascular disease (CVD) risk in primary and secondary prevention focus on the optimization of low-density lipoprotein-cholesterol (LDL-C) levels. As recommended in current guidelines for lowering blood cholesterol, statins in addition to lifestyle modifications remain the first-line therapy to reduce LDL-C in patients at CVD risk. However, despite optimal reduction of LDL-C with statins and, correction of other modifiable risk factors, CVD risk is not eliminated. The source of this residual risk may be due to other atherogenic lipid species such as reduced high-density lipoprotein cholesterol (HDL-C) and/or raised triglycerides (TG) which are only modestly affected by statin therapy.

The use of fibrates in the treatment of dyslipidaemia has changed significantly over recent years.

The potential of fibrate-statin combination treatment is discussed in guidelines and by the medical community. Fenofibrate treatment usually reduce TG by 40-50%, total cholesterol (TC) and LDL-C by 5-20%, as well as small dense LDL by 10-30%.

While fibrates are generally well tolerated, combination with a statin might increase the risk of side effects and potentially that of myopathy. In the ACCORD study, fenofibrate coadministered with simvastatin was neither associated with any increase in the incidence of myopathy over that observed with simvastatin monotherapy in patients with type 2 diabetes, nor pointing out any safety concerns for the coadministration.

In view of the demonstrated lipid benefit and good safety profile, fenofibrate is suitable for add-on therapy with a statin to minimize the CVD residual risk.

This post-marketing observational study is conducted to assess effectiveness of fenofibrate (145 mg daily) as adjuvant therapy to statins administered for 6 months in patients with hypertriglyceridemia and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Triglycerides level above 2,3 mmol/l.
* Patients having been prescribed fenofibrate 145 mg for at least 6 months AND who have been taking fenofibrate 145 mg no more than 3 days at the time of enrollment into the study.
* Patient who take statins at the time of enrollment into the study.
* Patients who have signed the informed consent to participate in this program.

Exclusion Criteria:

* Patients who took last dose within previous treatment course of fenofibrate less than 3 months ago.
* Statin-intolerant patients.
* Female patients during pregnancy or breastfeeding.
* diabetes mellitus (DM) type 1
* Participation in any other clinical or non-clinical study/program at present or within the latest 30 days.
* Patients with any other clinical states that make him/her ineligible for the program on the study doctor's opinion based on clinical assessment.
* Hepatic insufficiency (including biliary cirrhosis and unexplained persistent liver function abnormality).
* Known gallbladder disease.
* Severe chronic kidney disease (creatinine clearance <60 ml/min).
* Chronic or acute pancreatitis.
* Known photoallergy or phototoxic reaction during treatment with fibrates or ketoprofen.
* Hypersensitivity to the active substance(s) or to any of the excipients.
* Allergic to peanut or arachis oil or soya lecithin or related products due to risk of hypersensitivity reactions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The program will include adult patients with triglycerides > 2,3 mmol/l who are on statins and who are primary prescribed fenofibrate (or fenofibrate treatment break is at least 6 months) in accordance with ordinary physician practice in Russia.
  The decision to prescribe fenofibrate should be made not on the basis of this protocol but in accordance with the routine clinical practice and must be clearly separated from the decision to include the patient in the program. No additional diagnostic procedures (in addition to standard medical care) should be prescribed. The program included a questionnaire for patients to assess the quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Change of TG at Visit 3 (6 months of fenofibrate treatment) versus baseline level at Visit 1. | 6 months
  Triglycerides will be represented in mmol/L and change of TG will be displayed as mean difference of TG at Visit 3 vs. Visit 1.

SECONDARY OUTCOMES:
Change of LDL level at Visit 3 (6 months of fenofibrate treatment) versus baseline level at Visit 1 | 6months
  Low-density lipoproteins (LDL) will be represented in mmol/L and change of LDL will be displayed as mean difference of LDL at Visit 3 vs. Visit 1.
Change of lipid profile parameters (TC, HDL, non-HDL) at Visit 3 (6 months of fenofibrate treatment) versus baseline level at Visit 1 | 6 months
  Lipid profile includes total cholesterol (TC), high-density lipoproteins (HDL) and non-HDL. The lipid profile parameters will not be combined into 1 value and will be reported as separate values but results will be presented in the same unites of measure (mmol/L). Non-HDL is calculated as total cholesterol minus HDL cholesterol. Change of each lipid profile parameter will be displayed as mean difference of the result at Visit 3 vs. Visit 1.
Change of LDL level at Visit 2 (3 months of fenofibrate treatment) versus baseline level at Visit 1. | 3 months
  Low-density lipoproteins (LDL) will be represented in mmol/L and change of LDL will be displayed as mean difference of LDL at Visit 2 vs. Visit 1.
Change of lipid profile parameters (TC, TG, HDL, non-HDL) at Visit 2 (3 months of fenofibrate treatment) versus baseline level at Visit 1. | 3 months
  Lipid profile includes total cholesterol (TC), high-density lipoproteins (HDL) and non-HDL. The lipid profile parameters will not be combined into 1 value and will be reported as separate values but results will be presented in the same unites of measure (mmol/L). Non-HDL is calculated as total cholesterol minus HDL cholesterol. Change of each lipid profile parameter will be displayed as mean difference of the result at Visit 2 vs. Visit 1.
Change of C-reactive protein level at Visit 3 (6 months of fenofibrate treatment) versus baseline level at Visit 1 | 6 months
  Сhange of C-reactive protein (CRP) will be displayed as mean difference of CRP at Visit 3 vs. Visit 1.
Change of C-reactive protein level at Visit 2 (3 months of fenofibrate treatment) versus baseline level at Visit 1 | 3 months
  Сhange of C-reactive protein (CRP) will be displayed as mean difference of CRP at Visit 2 vs. Visit 1.
The average score on each of 8 scales of Short Form Survey Instrument (SF)-36 quality of life questionnaire at Visit 3 (6 months of fenofibrate treatment) versus baseline level at Visit 1. | 6 months
  The 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively, so that a high score defines a more favorable health state. Items in the same scale are averaged together to create the 8 scale scores.
  Patients will complete this self-reported questionnaire, containing 36 items, for evaluation of the quality of life after 6 months of treatment.
The average score on each of 8 scales of Short Form Survey Instrument (SF)-36 quality of life questionnaire at Visit 2 (3 months of fenofibrate treatment) versus baseline level at Visit 1 | 3 months
  The 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively, so that a high score defines a more favorable health state. Items in the same scale are averaged together to create the 8 scale scores.
  Patients will complete this self-reported questionnaire, containing 36 items, for evaluation of the quality of life after 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Solnyshkina, Study Director — Abbott
Locations (60):
- Russia (60):
  - City Polyclinic #14 (branch office), Barnaul
  - Clinical Diagnostic Centre, Bryansk
  - Polyclinic #1, Cheboksary
  - Diagnostic Centre, Cheboksary
  - Polyclinic #1, Chelyabinsk
  - Polyclinic, Chelyabinsk
  - Polyclinic #1, Irkutsk
  - Clinical hospital, Irkutsk
  - City Polyclinic #4, Irkutsk
  - Medical center, Kaliningrad
  - Polyclinic, Kazan'
  - Polyclinic #2 of Hospital #4, Kemerovo
  - Polyclinic, Kemerovo
  - City polyclinic 7/ ID 015, Krasnoyarsk
  - Dispensary, Krasnoyarsk
  - City Polyclinic #23, Moscow
  - City Polyclinic # 166 (branch office #2), Moscow
  - City Polyclinic #166 (branch office #3), Moscow
  - Clinical Diagnostic Centre #1 (branch office #4), Moscow
  - City Polyclinic #170 (branch office #2), Moscow
  - Medical center, Moscow
  - Polyclinic, Moscow
  - Regional hospital, Moscow Region
  - City Polyclinic, Moscow Region
  - Medical center, Moscow Region
  - Medical center, Nizhny Novgorod
  - Polyclinic #40, Nizhny Novgorod
  - Polyclinic of City Hospital #40, Nizhny Novgorod
  - Medical center, Nizhny Novgorod Region
  - Polyclinic, Nizhny Tagil
  - Polyclinic #4 ГКБ 6, Orenburg
  - Medical center, Perm
  - Clinical cardiologic dispensary, Perm
  - City Polyclinic #1 (branch office), Rostov-on-Don
  - City Polyclinic #7, Rostov-on-Don
  - City Polyclinic #1, Rostov-on-Don
  - Polyclinic of City Hospital #20, Rostov-on-Don
  - City Polyclinic #109, Saint Petersburg
  - City Polyclinic #116, Saint Petersburg
  - Medical unit, Saint Petersburg
  - City polyclinic #54 / ID 065, Saint Petersburg
  - City Polyclinic #71, Saint Petersburg
  - City Polyclinic #96, Saint Petersburg
  - Polyclinic #34, Saint Petersburg
  - City policlinic #3, Samara
  - Clinical hospital, Samara
  - Medical center, Samara
  - City Polyclinic #2, Saratov
  - Medical center, Smolensk
  - City hospital, Ufa
  - Polyclinic of City hospital #21, Ufa
  - Polyclinic # 2, Volgograd
  - City polyclinic 18 /ID 038, Volgograd
  - Polyclinic #30, Volgograd
  - Polyclinic #28, Volgograd
  - City Polyclinic #7, Voronezh
  - City hospital #4, Voronezh
  - Polyclinic, Yaroslavl
  - Polyclinic, Yekaterinburg
  - Medical center, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No